CLINICAL TRIAL: NCT04237584
Title: ESCALATE, A Phase III Randomized Study Comparing Enzalutamide or Darolutamide With Radium-223 vs Enzalutamide or Darolutamide With Placebo and the Effect Upon Symptomatic Skeletal Event-Free Survival for mCRPC Patients
Brief Title: A Study Comparing ARB With Radium-223 vs ARB Therapy With Placebo and the Effect Upon Survival for mCRPC Patients
Acronym: ESCALATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to insurmountable enrollment challenges affecting trial accrual, resulting from the rapidly evolving treatment options for advanced prostate cancer.
Sponsor: MANA RBM (Other)
Collaborators: Bayer (Industry); Carolina Urologic Research Center (Other); Tulane University (Other); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PC18-1005
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: mCRPC; ARB; Radiopharmaceutical
MeSH Terms: interventions — enzalutamide; radium Ra 223 dichloride; darolutamide

STUDY DESIGN:
Intervention Model Description: 12 week lead-in open-label androgen-receptor blocker (ARB) followed by up to 6 cycles of double-blind Radium-223 or placebo.
Who Masked: Participant, Investigator
Masking Description: Masking of Radium-223 or placebo only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Enzalutamide during Lead-in Period (Other): Randomized, open-label lead-in ARB (enzalutamide tablets, 160 mg PO QD) for 12 weeks.
  Interventions: Drug: Enzalutamide during Lead-in Period
- Lead-in Enzalutamide followed by Radium-223/Enzalutamide (Active Comparator): Randomized, open-label lead-in ARB (enzalutamide) for 12 weeks followed by randomized, double-blind Radium-223 IV at 55 kBq/kg IV up to 6 cycles (at 4 week intervals) with continued randomized open-label enzalutamide.
  Interventions: Drug: Lead-in Enzalutamide followed by Radium-223/Enzalutamide
- Lead-in Enzalutamide followed by Placebo/Enzalutamide (Placebo Comparator): Randomized, open-label lead-in ARB (enzalutamide) for 12 weeks followed by randomized, double-blind normal saline placebo IV up to 6 cycles (at 4 week intervals) with continued randomized open-label enzalutamide.
  Interventions: Drug: Lead-in Enzalutamide followed by Placebo/Enzalutamide
- Darolutamide during Lead-in Period (Other): Randomized, open-label lead-in ARB (darolutamide tablets, 300 mg PO BID) for 12 weeks.
  Interventions: Drug: Darolutamide during Lead-in Period
- Lead-in Darolutamide followed by Radium-223/Darolutamide (Active Comparator): Randomized, open-label lead-in ARB (darolutamide) for 12 weeks followed by randomized, double-blind Radium-223 IV at 55 kBq/kg IV up to 6 cycles (at 4 week intervals) with continued randomized open-label darolutamide.
  Interventions: Drug: Lead-in Darolutamide followed by Radium-223/Darolutamide
- Lead-in Darolutamide followed by Placebo/Darolutamide (Placebo Comparator): Randomized, open-label lead-in ARB (darolutamide) for 12 weeks followed by randomized, double-blind normal saline placebo IV up to 6 cycles (at 4 week intervals) with continued randomized open-label darolutamide.
  Interventions: Drug: Lead-in Darolutamide followed by Placebo/Darolutamide

INTERVENTIONS:
Drug: Enzalutamide during Lead-in Period — Participants will receive 12 weeks open-label lead-in ARB (enzalutamide) that will continue after double-blind randomization to radium-223 or placebo.
  Other Names: Xtandi
  Arms: Enzalutamide during Lead-in Period
Drug: Lead-in Enzalutamide followed by Radium-223/Enzalutamide — After a 12-week lead-in period of open-label enzalutamide, participants will be randomized to double-blind radium-223 or placebo. Participants will continue on their randomized, open-label enzalutamide.
  Other Names: Xofigo, Xtandi
  Arms: Lead-in Enzalutamide followed by Radium-223/Enzalutamide
Drug: Lead-in Enzalutamide followed by Placebo/Enzalutamide — After a 12-week lead-in period of open-label enzalutamide, participants will be randomized to double-blind radium-223 or placebo. Participants will continue on their randomized, open-label enzalutamide.
  Other Names: Placebo, Xtandi
  Arms: Lead-in Enzalutamide followed by Placebo/Enzalutamide
Drug: Darolutamide during Lead-in Period — Participants will receive 12 weeks open-label lead-in darolutamide that will continue after double-blind randomization to radium-223 or placebo.
  Other Names: Nubeqa
  Arms: Darolutamide during Lead-in Period
Drug: Lead-in Darolutamide followed by Radium-223/Darolutamide — After a 12-week lead-in period of open-label darolutamide, participants will be randomized to double-blind radium-223 or placebo. Participants will continue on their randomized, open-label darolutamide.
  Other Names: Xofigo, Nubeqa
  Arms: Lead-in Darolutamide followed by Radium-223/Darolutamide
Drug: Lead-in Darolutamide followed by Placebo/Darolutamide — After a 12-week lead-in period of open-label darolutamide, participants will be randomized to double-blind radium-223 or placebo. Participants will continue on their randomized, open-label darolutamide.
  Other Names: Placebo, Nubeqa
  Arms: Lead-in Darolutamide followed by Placebo/Darolutamide

SUMMARY:
This is a randomized, multi-center, double-blind, Phase III study of radium-223 plus enzalutamide or darolutamide compared to enzalutamide or darolutamide treatment plus placebo.

DETAILED DESCRIPTION:
The hypothesis investigators will test in this study is whether layering radium-223 following 16 weeks of enzalutamide or darolutamide exposure in patients demonstrating a biochemical response improves disease outcomes. By adding radium-223 following a potential bone flare phenomenon [after first 12-14 weeks of therapy with an androgen receptor blocker (ARB)], including patients expected to have durable response to systemic therapy, and mandating the use of bone protective agents during treatment, the investigators aim to demonstrate an optimal time to add radium-223 in the mCRPC landscape.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent.
2. Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma.
3. Men ≥ 18 years.
4. ECOG performance status of 0 or 1 at screening.
5. Metastatic to bone with ≥ 2 bone metastases (area of increased uptake on 99mTc bone scan); equivocal lesions on the bone scan must be confirmed by standard X-ray, CT, or MRI.
6. Patients must have progressive metastatic castration-resistant prostate cancer (mCRPC) at screening and on androgen deprivation therapy (ADT) as evidenced by either:

   1. For patients who manifest disease progression solely as a rising prostate-specific antigen (PSA) level - documentation of a sequence of two rising PSA values at a minimum of 1-week apart with the Screening value ≥1 ng/ml (see Appendix D);
   2. For patients with disease progression manifested in the bone, irrespective of progression by rising PSA - defined by the appearance of 2 or more new skeletal lesions demonstrated by 99Tc bone imaging. Ambiguous results should be confirmed by other imaging modalities than bone scan and x-ray (e.g.: CT-scan or MRI).
   3. For patients with disease progression manifested at nodal sites, irrespective of progression by rising PSA - progression defined per RECIST 1.1.
7. Ongoing ADT with luteinizing hormone-releasing hormone (LHRH) agonist or antagonist or bilateral orchiectomy.
8. Use of bone health agents (denosumab or zoledronic acid or other bisphosphonates) starting any time prior to R1 unless contraindicated or considered not in the best interest of the patient. A waiver must be approved by the medical monitor if bone health agents cannot be used. Bone health agents should be continued throughout both RT1 and RT2 treatment periods.
9. Adequate bone marrow and organ function as defined by:

   1. Hemoglobin ≥ 10.0 g/dL
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. Platelets ≥ 100 x 109/L
   4. Serum creatinine ≤ 1.95 mg/dL
   5. Estimated creatinine clearance >/= 30 mL/min by Cockroft-Gault calculation
   6. Alanine aminotransferase (ALT) ≤ 175 U/L
   7. Aspartate aminotransferase (AST) ≤ 100 U/L
   8. Total bilirubin ≤ 1.8 mg/dL (unless the patient a diagnosis of Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin; in patients with Gilbert's, the total bilirubin should be less than 6 mg/dL if patient has Gilbert's and the elevation should be seen in the unconjugated or indirect bilirubin measurement)
   9. LDH ≤ 224 U/L at screening.
   10. Albumin ≥ 2.5 g/dL
10. Fertile male patients, defined as all males physiologically capable of conceiving offspring with female partners of child-bearing potential, must be willing to use condoms plus spermicidal agent during the study treatment period and for 6 months after the last dose of study drug, and not father a child or donate sperm during this period.
11. The treating site investigator deems RT1 (Enzalutamide or Darolutamide) treatment safe and feasible.

    Subjects must meet the remaining inclusion criteria in order to be qualified for the second randomization (R2). Only subjects that complete the initial 12 weeks of run-in RT1 should be evaluated. Prior inclusion criteria do not need to be re-evaluated:
12. Patients must have a documented ≥ 30% decline of PSA at any time during the 12 weeks of RT1.
13. Patients must have no evidence of visceral metastatic disease at the time of RT2 randomization
14. Ongoing treatment with RT1 and bone health agents at time of RT2 randomization.
15. The treating site investigator deems RT2 (Ra-223 dichloride) treatment safe and feasible.

Exclusion Criteria:

1. Pathological finding consistent with small cell carcinoma of the prostate.
2. Prior chemotherapy for CRPC. Prior docetaxel for hormone-sensitive disease is permitted under the following conditions: started within 3 months of ADT initiation, given for a maximum of 6 cycles and progression occurred > 6 months after the last dose of docetaxel.
3. Prior treatment for mCRPC or CRPC. However, the following therapies are permitted and not exclusionary: Sipuleucel-T, 5-alpha-reductase inhibitors, estrogens, or older antiandrogens (such as flutamide, bicalutamide, or nilutamide).
4. Prior treatment for more than 2 months with CYP17 inhibitors (e.g. abiraterone or orteronel).
5. Prior treatment for more than 2 months with agents inhibiting androgen receptor signaling (e.g. enzalutamide, apalutamide, or darolutamide).
6. Prior hemibody or whole-body external radiotherapy. Other types of prior external radiotherapy and brachytherapies are allowed.
7. Prior therapy with radionuclides (e.g., radium-223, strontium-89, samarium-153, rhenium-186, rhenium-188, actinium-225 and lutetium-177).
8. Current involvement in any drug or device trial involving investigational agent or medical device within the last 28 days prior to R1.
9. In general, any prior investigational agent for nmCRPC/mCRPC; however, may be reviewed by medical monitor/PIs for waiver consideration, on a case-by-case basis.
10. Hypersensitivity to compounds related to enzalutamide, darolutamide, or Ra-223.
11. A blood transfusion ≤ 28 days prior to R1.
12. Major surgical procedures ≤ 28 days or minor surgical procedures ≤7 days prior to R1. No waiting period is required following port-a-cath placement.
13. Patients with visceral metastases, clinical evidence of central nervous system metastases, or leptomeningeal tumor spread as demonstrated via CT/MRI of chest, abdomen, pelvis, and CNS (if needed). CT/MRI of the CNS only performed if suspicion of CNS metastases or leptomeningeal tumor spread. Nodules < 1 cm alone will not be considered visceral metastases. Renal masses < 3 cm will not be considered exclusionary.
14. Serious active infection at the time of screening or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
15. Presence of other active cancers, or history of treatment for invasive cancer ≤2 years of R1. Patients with Stage I/II cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) and superficial bladder cancer are eligible, as are patients with history of non-melanoma skin cancer.
16. Any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shore, MD, Study Chair — Carolina Urologic Research Center
Locations (1):
- Research Site, Myrtle Beach, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from Jun 2020- Jul 2021 at selected medical centers that specialized in the treatment of advanced prostate cancer.
Pre-assignment Details: 23 subjects signed ICF. 2/23 subjects screen failed without reporting any adverse events and received no study treatments. 21/23 subjects signing ICF met all entry criteria and were randomized to Lead-in ARB (R1). 5 subjects discontinued the study during Lead-in ARB. Although 16 subjects randomized to R2, 2 of the subjects randomized to Enzalutamide + Placebo did not receive any cycles due to the early termination of the study and are reported only in the Lead-in Enzalutamide safety group.
Groups:
- Enzalutamide + Ra-223: Lead-in Enzalutamide 12 weeks followed by Ra-223 up to 6 cycles (at 4 week intervals) with continued Enzalutamide.
- Darolutamide + Ra-223: Lead-in Darolutamide 12 weeks followed by Ra-223 up to 6 cycles (at 4 week intervals) with continued Darolutamide.
- Enzalutamide + Placebo: Lead-in Enzalutamide 12 weeks followed by Placebo (normal saline) up to 6 cycles (at 4 week intervals) with continued Enzalutamide.
- Darolutamide + Placebo: Lead-in Darolutamide 12 weeks followed by Placebo (normal saline) up to 6 cycles (at 4 week intervals) with continued Darolutamide.
Period: R1- Lead-in ARB Treatment (12 Weeks)
Arm/Group | Enzalutamide + Ra-223 | Darolutamide + Ra-223 | Enzalutamide + Placebo | Darolutamide + Placebo
Started | 5 | 5 | 6 | 5
Completed | 4 | 4 | 3 | 3
Not Completed | 1 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Did not meet R2 entry criteria | 1 | 1 | 0 | 1
Not completed — Randomized R2 (no cycles given) | 0 | 0 | 2 | 0
Period: R2- ARB Treatment With Ra-223 or Placebo
Arm/Group | Enzalutamide + Ra-223 | Darolutamide + Ra-223 | Enzalutamide + Placebo | Darolutamide + Placebo
Started | 4 | 4 | 3 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 3 | 3
Not completed — Sponsor Decision | 4 | 4 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lead-in Enzalutamide Followed by Radium-223/Enzalutamide: 12-week lead-in of open-label Enzalutamide followed by radium-223. Participants continued on their randomized, open-label Enzalutamide.
- Lead-in Darolutamide Followed by Radium-223/Darolutamide: 12-week lead-in of open-label Darolutamide followed by radium-223. Participants continued on their randomized, open-label Darolutamide.
- Lead-in Enzalutamide Followed by Placebo/Enzalutamide: 12-week lead-in of open-label Enzalutamide followed by placebo. Participants continued on their randomized, open-label Enzalutamide.
- Lead-in Darolutamide Followed by Placebo/Darolutamide: 12-week lead-in of open-label Darolutamide followed by placebo. Participants continued on their randomized, open-label Darolutamide.
- Total: Total of all reporting groups
Arm/Group | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide | Total
Number analyzed (Participants) | 5 | 5 | 6 | 5 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 1 | 1
  >=65 years | 5 | 5 | 6 | 4 | 20
Sex/Gender, Customized [Number; unit: participants]
  Males | 5 | 5 | 6 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 4 | 6 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 5 | 4 | 5 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 6 | 5 | 21
Concomitant use of bone health agents (osteoclast inhibitors) [Count of Participants; unit: Participants] | 5 | 5 | 6 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Skeletal Event-free Survival (SSE-FS)
Description: SSE-FS is a composite endpoint, composed of 4 events that indicate disease progression:
  * the first use of external-beam radiation therapy to relieve skeletal tumor-related symptoms
  * the occurrence of new symptomatic pathologic bone fractures.
  * the occurrence of new symptomatic spinal cord compression
  * a tumor-related orthopedic surgical intervention
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects that met primary endpoint (occurrence of SSE-FS).
Measure: Count of Participants; unit: Participants
Groups:
- Lead-in Enzalutamide Only (no Cycles): Lead-in Enzalutamide only. No Cycles.
- Lead-in Darolutamide Only (no Cycles): Lead-in Darolutamide only. No Cycles.
- Lead-in Enzalutamide Followed by Radium-223/Enzalutamide: Randomized, Open-label Lead-in ARB (enzalutamide) followed by Radium-223 + Enzalutamide.
- Lead-in Darolutamide Followed by Radium-223/Darolutamide: Randomized, Open-label Lead-in ARB (darolutamide) followed by Radium-223 + Darolutamide.
- Lead-in Enzalutamide Followed by Placebo/Enzalutamide: Randomized, Open-label Lead-in ARB (enzalutamide) followed by Placebo + Enzalutamide.
- Lead-in Darolutamide Followed by Placebo/Darolutamide: Randomized, Open-label Lead-in ARB (darolutamide) followed by Placebo + Darolutamide.
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 2 | 1

2. Secondary Outcome: Overall Survival (OS)
Description: Number of subjects who survived between RT2 randomization through data cut-off.
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects with who survived.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 4 | 3 | 4 | 4 | 3 | 3

3. Secondary Outcome: Time to Chemotherapy Initiation
Description: Number of subjects who began docetaxel or cabazitaxel treatment during the study.
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects who started docetaxel or cabazitaxel treatment during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Number of subjects with bone scan progression per PCWG3 criteria, and/or progression by CT/MRI per RECIST 1.1 criteria, or death from any cause following RT2. Radiological progression is interpreted by local assessment only.
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects who experienced radiological progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 1 | 1

5. Secondary Outcome: Safety Profile of Androgen Receptor Blocker (ARB) Therapy With or Without Radium-223.
Description: Safety profile of androgen receptor blockers (enzalutamide or darolutamide) with or without radium-223; number of participants with treatment-related adverse events as assessed by CTCAE v5.0. Reported only in the AE reporting module.
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects followed for safety. Safety data reported in AE section.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 3 | 3
Participants | 4 | 2 | 4 | 4 | 3 | 3

6. Secondary Outcome: Occurrence of AESI: Bone Fractures (Pathologic and Non-pathologic)
Description: Assess occurrence of AESI: fractures (pathologic and non-pathologic).
Time Frame: approximately 1 year and 8 months
Population: No analysis was performed. Outcome measure includes only number (%) of subjects with AESI.
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Enzalutamide Only (no Cycles) | Lead-in Darolutamide Only (no Cycles) | Lead-in Enzalutamide Followed by Radium-223/Enzalutamide | Lead-in Darolutamide Followed by Radium-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
Number analyzed (Participants) | 11 | 10 | 4 | 4 | 3 | 3
Participants | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection started at the time each subject signed informed consent and continued to be collected until each subject was 30 days post-last dose of study medication (enzalutamide, darolutamide, Ra-223, or placebo). The duration of the study was approximately 1 year and 8 months.
Groups:
- 12 Weeks Lead-in Enzalutamide Only (No Cycles): 12 weeks of Lead-in Enzalutamide without any cycles
- 12 Weeks Lead-in Darolutamide Only (No Cycles): 12 weeks of Lead-in Darolutamide without any cycles
- Lead-in Enzalutamide Followed by Ra-223/Enzalutamide: 12 weeks Lead-in Enzalutamide followed by up to 6 (once monthly) Ra-223 cycles + continued Enzalutamide
- Lead-in Darolutamide Followed by Ra-223/Darolutamide: 12 weeks Lead-in Darolutamide followed by up to 6 (once monthly) Ra-223 cycles + continued Darolutamide
- Lead-in Enzalutamide Followed by Placebo/Enzalutamide: 12 weeks Lead-in Enzalutamide followed by up to 6 (once monthly) Placebo cycles + continued Enzalutamide
- Lead-in Darolutamide Followed by Placebo/Darolutamide: 12 weeks Lead-in Darolutamide followed by up to 6 (once monthly) Placebo cycles + continued Darolutamide
Arm/Group | 12 Weeks Lead-in Enzalutamide Only (No Cycles) | 12 Weeks Lead-in Darolutamide Only (No Cycles) | Lead-in Enzalutamide Followed by Ra-223/Enzalutamide | Lead-in Darolutamide Followed by Ra-223/Darolutamide | Lead-in Enzalutamide Followed by Placebo/Enzalutamide | Lead-in Darolutamide Followed by Placebo/Darolutamide
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 1/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 4/4 | 4/4 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Weeks Lead-in Enzalutamide Only (No Cycles) (N=4) | 12 Weeks Lead-in Darolutamide Only (No Cycles) (N=3) | Lead-in Enzalutamide Followed by Ra-223/Enzalutamide (N=4) | Lead-in Darolutamide Followed by Ra-223/Darolutamide (N=4) | Lead-in Enzalutamide Followed by Placebo/Enzalutamide (N=3) | Lead-in Darolutamide Followed by Placebo/Darolutamide (N=3)
Syncope (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — SAE was not attributable to study treatments
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — SAE was not attributable to study treatments
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — SAE was not attributable to study treatments
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — SAE was not attributable to study treatments
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Weeks Lead-in Enzalutamide Only (No Cycles) (N=4) | 12 Weeks Lead-in Darolutamide Only (No Cycles) (N=3) | Lead-in Enzalutamide Followed by Ra-223/Enzalutamide (N=4) | Lead-in Darolutamide Followed by Ra-223/Darolutamide (N=4) | Lead-in Enzalutamide Followed by Placebo/Enzalutamide (N=3) | Lead-in Darolutamide Followed by Placebo/Darolutamide (N=3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Confusional state (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
ESCALATE (PC18-1005) was terminated early due to enrollment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT04237584/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04237584/ICF_001.pdf